CLINICAL TRIAL: NCT04622007
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Tomivosertib in Combination With Anti-PD-(L)1 Therapy in Subjects With NSCLC as First Line Therapy or When Progressing on Single-Agent First-Line Anti PD (L)1 Therapy
Brief Title: Tomivosertib Combined With Pembrolizumab in Subjects With PD-L1 Positive NSCLC (KICKSTART)
Acronym: KICKSTART
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Effector Therapeutics (Industry)
Collaborators: Medpace, Inc. (Industry); ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: eFT508-0011
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tomivosertib; pembrolizumab; Pemetrexed

STUDY DESIGN:
Intervention Model Description: In each Cohort approximately 60 eligible Subjects were targeted to be randomized to receive tomivosertib or matching placebo in combination with pembrolizumab (and pemetrexed, Cohort C). Cohorts A and C were closed to enrollment early due to recruitment challenges. In Cohort B, 54 subjects received blinded IP (tomivosertib or matching placebo) in combination with pembrolizumab as first line therapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In all cohorts, investigational product (IP, tomivosertib or placebo) will be blinded and pembrolizumab will be open label. On Cohort C, pembrolizumab and pemetrexed will be open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- A1 Tomi + Current Pembro (Experimental): Subjects who have initiated pembrolizumab as a single agent and in accordance with the package insert will receive tomivosertib in addition to pembrolizumab.
  Interventions: Drug: Tomivosertib; Biological: Pembrolizumab
- Pbo + Current Pembro (Placebo Comparator): Subjects who have initiated pembrolizumab as a single agent and in accordance with the package insert, will receive matching placebo in addition to pembrolizumab.
  Interventions: Biological: Pembrolizumab
- B1 Tomi + Pembro (Experimental): Subjects will initiate pembrolizumab as first-line therapy and receive tomivosertib.
  Interventions: Drug: Tomivosertib; Biological: Pembrolizumab
- Pbo + Pembro (Placebo Comparator): Subjects will initiate pembrolizumab as first-line therapy and receive matching placebo.
  Interventions: Biological: Pembrolizumab
- C1 Tomi + Pembro + Pemetrexed (Non-sqamous) or Tomi + Pembro (Squamous) (Experimental): Subjects who have completed 4 to 6 cycles of platinum-based chemotherapy doublet will receive tomi plus pembrolizumab and pemetrexed (non-squamous NSCLC) or tomi plus pembro as a single agent (squamous) in accordance with the package insert.
  Interventions: Drug: Tomivosertib; Biological: Pembrolizumab; Drug: Pemetrexed
- Pbo + Pembro + Pemetrexed (Non-sqamous) or Pbo + Pembro (Squamous) (Placebo Comparator): Subjects who have completed 4 to 6 cycles of platinum-based chemotherapy doublet will receive placebo plus pembrolizumab and pemetrexed (non-squamous NSCLC) or placebo plus pembro as a single agent (squamous) in accordance with the package insert.
  Interventions: Biological: Pembrolizumab; Drug: Pemetrexed

INTERVENTIONS:
Drug: Tomivosertib — Tomivosertib (eFT508) will be taken at 100 mg twice daily (bid) with meals
  Other Names: eFT508
  Arms: A1 Tomi + Current Pembro; B1 Tomi + Pembro; C1 Tomi + Pembro + Pemetrexed (Non-sqamous) or Tomi + Pembro (Squamous)
Biological: Pembrolizumab — Subjects will initiate or continue to receive pembrolizumab at either 200 mg intravenously (IV) at a frequency of every 3 weeks or 400 mg IV at a frequency of every 6 weeks.
  Other Names: Keytruda®
Drug: Pemetrexed — Subjects will initiate pemetrexed at 500 mg/m2 intravenously (IV) at a frequency of every 3 weeks.
  Other Names: Alimta®
  Arms: C1 Tomi + Pembro + Pemetrexed (Non-sqamous) or Tomi + Pembro (Squamous); Pbo + Pembro + Pemetrexed (Non-sqamous) or Pbo + Pembro (Squamous)

SUMMARY:
Tomivosertib combined with pembrolizumab in Subjects with PD-L1 positive NSCLC

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled Trial of Tomivosertib in Combination With Anti-PD-(L)1 Therapy in Subjects With Non-Small Cell Lung Cancer as First Line Therapy or When Progressing on Single-Agent First-Line Anti PD (L)1 Therapy

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Cohort A: Subjects who meet all of the following criteria will be eligible to participate in Cohort A of the study:

1. Have initiated first-line therapy for NSCLC with pembrolizumab and satisfy the following:

* Have tumor PD-L1 ≥1% by 22C3 IHC;
* Are judged by the Principal Investigator as tolerating pembrolizumab monotherapy; and
* Have been on pembrolizumab for at least 3 months (measured from actual first dose date to first dose date of the current study) and the most recent scans are the first scans to objectively demonstrate Progressive Disease per RECIST 1.1
* The first scan conducted a minimum of 21 days after first dose of anti-PD-(L)1 therapy must have shown either SD, PR, or CR (ie, not Progressive Disease) per RECIST 1.1; and
* The 2 most recent scans (including 1 demonstrating Progressive Disease) are available to be reviewed

Inclusion Criterion for Cohort B

Subjects who meet the following criterion will be eligible to participate in Cohort B of the study:

1. Are eligible for single-agent pembrolizumab for advanced/metastatic NSCLC in accordance with the package insert and have tumor PD-L1 ≥50% by 22C3 IHC

• Must not have been treated previously with platinum-based chemotherapy in the advanced/metastatic setting. Note: Subjects may have received chemotherapy and/or anti PD (L)1 therapy in the neo/adjuvant setting, provided the last dose of therapy was >9 months prior to randomization.

All cohorts require PD-L1 testing (TPS as determined by an FDA-approved test: subjects in Cohort B must specifically have PD-L1 testing using the PD-L1 IHC 22C3 pharmDx test kit). Subjects in Cohort B for whom PD-L1 testing was not performed with the required IHC 22C3 pharmDx test kit may be randomized if all other study criteria have been met, pending retest with the required IHC 22C3 pharmDx test kit.

Subjects who meet the following criterion will be eligible to participate in Cohort C of the study:

1. Have initiated IL therapy for NSCLC and completed all planned (eg, 4 to 6 cycles) platinum-based chemotherapy with at least 2 cycles in combination with pembrolizumab; must not have had progressive disease on tumor staging imaging scans following completion of all planned platinum chemotherapy

* Are eligible for maintenance therapy with pembrolizumab ± pemetrexed in accordance with the package insert
* Have tumor PD-L1 ≥1%
* The last dose of platinum-based chemotherapy must be within 8 weeks of the first dose of the study drug in this study

Inclusion Criterion for All Cohorts

* Subjects must also meet all of the following criteria to be eligible to participate in the study:

  1. Have histologically confirmed NSCLC that is inoperable, locally advanced or metastatic (Stage IIIb/IV)
  2. Have available at the site a representative formalin-fixed, paraffin-embedded tumor specimen that enabled diagnosis of NSCLC in a tissue block (preferred) or 10 unstained, serial slides, accompanied by an associated pathology report. Note: If the archival tissue is neither sufficient nor available, the subject may still be eligible, upon discussion with the Medical Monitor
  3. Have provided written informed consent and any authorizations required by local law
  4. Are ≥18 years of age
  5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

1. Have NSCLC with epidermal growth factor receptor or anaplastic lymphoma kinase genomic tumor aberrations
2. Have gastrointestinal (GI) disease (eg, gastric or intestinal bypass surgery, pancreatic enzyme insufficiency, malabsorption syndrome, symptomatic inflammatory bowel disease, chronic diarrheal illness, and/or bowel obstruction) that may interfere with drug absorption or with interpretation of GI AEs
3. Have known symptomatic brain metastases requiring >10 mg/day of prednisone (or its equivalent). Subjects with previously diagnosed brain metastases are eligible if they have completed their treatment, have recovered from the acute effects of radiation therapy or surgery prior to randomization, fulfill the steroid requirement for these metastases, the 2 most recent serial magnetic resonance imaging (MRI) scans conducted >28 days apart show no central nervous system progression, and are neurologically stable and asymptomatic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2024-10-14 (Estimated); Study Completion 2024-12-09 (Estimated)

PRIMARY OUTCOMES:
To characterize the progression-free survival (PFS) of tomivosertib when added to pembrolizumab as a first-line treatment; and | 2 years
  Defined as the time from randomization to the first occurrence of disease progression as assessed by the Investigator using RECIST 1.1 or death from any cause, whichever occurs earlier.
To characterize the PFS of tomivosertib when added to pembrolizumab as first line therapy. | 2 years
  Defined as the time from randomization to the first occurrence of disease progression as assessed by the Investigator using RECIST 1.1 or death from any cause, whichever occurs earlier.
To characterize the PFS of tomivosertib when added to pembrolizumab and pemetrexed in non-squamous NSCLC, and pembrolizumab in squamous NSCLC as first line maintenance therapy. | 2 years
  Defined as the time from randomization to the first occurrence of disease progression as assessed by the Investigator using RECIST 1.1 or death from any cause, whichever occurs earlier.

SECONDARY OUTCOMES:
To characterize the PFS of tomivosertib when added to pembrolizumab in Cohorts A, B, and B C individually and combined | 2 years
  Defined as the time from randomization to the first occurrence of disease progression as assessed by the Investigator using RECIST 1.1 or death from any cause, whichever occurs earlier.
To characterize the PFS of tomivosertib when added to pembrolizumab as a first-line treatment in subjects with NSCLC | 2 years
  Defined as the time from randomization to the first occurrence of disease progression as assessed by the Investigator using RECIST 1.1 or death from any cause, whichever occurs earlier. Objective response per RECIST 1.1, as assessed by the BIRC.
To characterize the PFS of tomivosertib when added to pembrolizumab and pemetrexed in non-squamous NSCLC, and pembrolizumab in squamous NSCLC as a first-line maintenance treatment in subjects with NSCLC. | 2 years
  Defined as the time from randomization to the first occurrence of disease progression as assessed by the Investigator using RECIST 1.1 or death from any cause, whichever occurs earlier. Objective response per RECIST 1.1, as assessed by the BIRC.
To characterize the PFS of tomivosertib when added to pembrolizumab after first radiographic progression on pembrolizumab monotherapy | 2 years
  Defined as the time from randomization to the first occurrence of disease progression as assessed by the Investigator using RECIST 1.1 or death from any cause, whichever occurs earlier. Objective response per RECIST 1.1, as assessed by the BIRC

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Warner, MD, Study Director — EFFECTOR Therapeutics, Inc.
Locations (144):
- United States (131):
  - Southern Cancer Center, Daphne, Alabama
  - Southern Cancer Center, PC (Mobile Infirmary Circle), Mobile, Alabama
  - Southern Cancer Center, PC (Airport Blvd), Mobile, Alabama
  - Southern Cancer Center, PC (Dauphin St), Mobile, Alabama
  - Arizona Oncology Associates, PC - HAL (W Bell Rd), Glendale, Arizona
  - Arizona Oncology Associates, PC - NAHOA (W. McDowell), Goodyear, Arizona
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Arizona Oncology Associates, PC-NAHOA (N. Windsong), Prescott Valley, Arizona
  - Arizona Oncology Associates (N. Pima Rd), Scottsdale, Arizona
  - Arizona Oncology Associates, PC - HAL, Scottsdale, Arizona
  - Arizona Oncology Associates, PC - HAL, Tempe, Arizona
  - Arizona Oncology Associates, PC - HOPE (W. Orange Grove), Tucson, Arizona
  - Arizona Oncology Associates, PC - HOPE (W. Rudasill Rd), Tucson, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Arizona Oncology Associates, PC - HOPE (West St.), Tucson, Arizona
  - University of California, Los Angeles (UCLA) - Alhambra, Alhambra, California
  - Comprehensive Blood And Cancer Center, Bakersfield, California
  - TOI Clincal Research, Cerritos, California
  - California Cancer Associates for Research & Excellence (San Diego Pacific Oncology and Hematology Associates) - Encinitas, Encinitas, California
  - City of Hope - Long Beach Elm, Long Beach, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Mercy Cancer Center, Merced, California
  - Mercy UC Davis Center Center, Merced, California
  - Keck Medicine of USC Norris Oncology/Hematology, Newport Beach, California
  - University of California - Irvine Medical Center, Orange, California
  - University of California, Los Angeles (UCLA) - Porter Ranch, Porter Ranch, California
  - St. Mary's Medical Center - San Francisco, San Francisco, California
  - Dignity Health- SLO Oncology and Hematology, San Luis Obispo, California
  - University of California, Los Angeles (UCLA) - San Luis Obispo, San Luis Obispo, California
  - California Cancer Associates for Research & Excellence (San Diego Pacific Oncology and Hematology Associates) - San Marcos Cancer Center, San Marcos, California
  - Mission Hope Cancer Center, Santa Maria, California
  - Dignity Health St. Joseph's Medical Center Stockton, Stockton, California
  - Stockton Hematology Oncology Medical Group (Stockton), Stockton, California
  - Santa Clarita - UCLA, Valencia, California
  - Ventura - UCLA, Ventura, California
  - PIH Health Hospital - Whittier, Whittier, California
  - Rocky Mountain Cancer Centers (South Potomac St), Aurora, Colorado
  - Rocky Mountain Cancer Centers (Arapahoe Ave), Boulder, Colorado
  - Rocky Mountain Cancer Centers (E Arapahoe Rd), Centennial, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs CO (Peregrine), Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers (Williams St), Denver, Colorado
  - Rocky Mountain Cancer Centers (E. Hale Parkway), Denver, Colorado
  - Rocky Mountain Cancer Centers (West 2nd Place), Lakewood, Colorado
  - Rocky Mountain Cancer Centers (W Dry Creek Circle), Littleton, Colorado
  - Rocky Mountain Cancer Centers (Ridge Gate Parkway), Lone Tree, Colorado
  - Rocky Mountain Cancer Centers (E. Ken Pratt Blvd), Longmont, Colorado
  - Rocky Mountain Cancer Centers (Ridge Gate Parkway), Pueblo, Colorado
  - Rocky Mountain Cancer Centers (Huron St), Thornton, Colorado
  - ASCLEPES Research Centers, Brooksville, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Cancer Care Centers of Brevard (Melbourne), Melbourne, Florida
  - University of Florida (UF) Health Cancer Center - Orlando Health, Orlando, Florida
  - Cancer Care Centers of Brevard, Palm Bay, Florida
  - Memorial Cancer Institute at Memorial West Hospital, Pembroke Pines, Florida
  - Woodlands Medical Specialists, PA, Pensacola, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Baptist Health - Lexington, Lexington, Kentucky
  - Baptist Health - Louisville, Louisville, Kentucky
  - Luminus Health Research Institute, Inc., Annapolis, Maryland
  - Maryland Oncology Hematology, P.A. (Rockledge Dr), Bethesda, Maryland
  - Maryland Oncology Hematology, P.A. (Matapeake Business Dr), Brandywine, Maryland
  - Maryland Oncology Hematology, P.A. (Woodyard Rd), Clinton, Maryland
  - Maryland Oncology Hematology, P.A, Columbia, Maryland
  - Maryland Oncology Hematology, P.A. (Thomas Johnson Dr), Frederick, Maryland
  - Maryland Oncology Hematology, P.A. (Good Luck Rd), Lanham, Maryland
  - Maryland Oncology Hematology, P.A. (Medical Center Drive), Rockville, Maryland
  - Maryland Oncology Hematology, P.A. (Healing Way), Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Metro Minnesota CCOP, Saint Louis Park, Minnesota
  - Mercy Cancer Center, Joplin, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Broome Oncology, Binghamton, New York
  - Broome Oncology, LLC (Harrison St), Johnson City, New York
  - Columbia University Medical Center, New York, New York
  - Columbia University, New York, New York
  - Messino Cancer Center, Asheville, North Carolina
  - Mercy Hematology and Oncology Associates, Canton, Ohio
  - Gabrail Cancer Center, Canton, Ohio
  - VA Medical Center- Dayton, Dayton, Ohio
  - Tri-County Hematology & Oncology Associates, Dover, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Tri-County Hematology & Oncology Associates - Massillon, Massillon, Ohio
  - University of Toledo, Toledo, Ohio
  - Willamette Valley Cancer Institute and Research Ctr, Eugene, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Prairie Lakes Cancer Center, Watertown, South Dakota
  - Texas Oncology - West Texas (Antilley Rd), Abilene, Texas
  - Texas Oncology-Austin Midtown (W. 38th St), Austin, Texas
  - Texas Oncology-Austin Central (Balcones Dr.), Austin, Texas
  - Texas Oncology - South Austin, Austin, Texas
  - Texas Oncology Gulf Coast - Beaumont (College St), Beaumont, Texas
  - Texas Oncology Gulf Coast - Beaumont Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology-Carrollton (N Josey Lane), Carlton, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Denton, Denton, Texas
  - Texas Oncology - West Texas (Grandview Ave), El Paso, Texas
  - Texas Oncology - West Texas, El Paso, Texas
  - Texas Oncology - West Texas (Gateway Blvd E), El Paso, Texas
  - Texas Oncology - West Texas (Joe Battle Dr), El Paso, Texas
  - Texas Oncology - Flower Mound - Carrollton, Flower Mound, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology-Grapevine, Grapevine, Texas
  - Valley Cancer Associates, Harlingen, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - Texas Oncology Gulf Coast (Willowbrook), Houston, Texas
  - Texas Oncology - Longview Cancer Center, Longview, Texas
  - Texas Oncology - West Texas (Odessa), Odessa, Texas
  - Texas Oncology - Palestine, Palestine, Texas
  - Texas Oncology - Paris, Paris, Texas
  - Texas Oncology - Plano East, Plano, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Texas Oncology - Waco, Waco, Texas
  - Texas Oncology Golf Coast - Deke Slayton Cancer Center, Webster, Texas
  - Virginia Cancer Specialists, PC (Kenmore Ave), Alexandria, Virginia
  - Virginia Cancer Specialists, PC (N George Mason Dr), Arlington, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Cancer Specialists, PC (Lake Manassas Dr), Gainesville, Virginia
  - Virginia Cancer Specialists, PC (Riverside Pkwy), Leesburg, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
  - MultiCare Regional Cancer Center, Spokane, Washington
  - West Virginia University Cancer Institute, Morgantown, West Virginia
- Australia (3):
  - Gold Coast Cancer Care - Pindara, Benowa, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Ballarat Regional Integrated Cancer Center, Ballarat, Victoria
- Georgia (10):
  - High Technology Hospital MedCenter Ltd, Batumi, Adjara
  - TIM - Tbilisi Institute of Medicine LLC, Tbilisi, Tbilisa
  - JSC Vian - Kutaisi Referral Hospital, Kutaisi
  - Israel-Georgia Medical Research Clinic Healthycore LLC, Tbilisi
  - Todua Clinic LLC, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic LLC, Tbilisi
  - Oncology Scientific Research Center LLC, Tbilisi
  - Multiprofile Clinic Consilium Medulla LLC, Tbilisi
  - JSC Viani, Tbilisi
  - Caucasus Medical Centre LLC, Tbilisi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo H, Huang S. Inhibition of MNK pathway sensitizes nasopharyngeal carcinoma to radiotherapy. Anticancer Drugs. 2024 Feb 1;35(2):155-162. doi: 10.1097/CAD.0000000000001542. Epub 2023 Sep 11. PMID 37694854